CLINICAL TRIAL: NCT01232985
Title: An Open-Label Pilot Study to Determine the Efficacy and Tolerability of a Device, RD047-26 for the Treatment of Mild to Moderate Atopic Dermatitis With Associated Pruritus in Adults
Brief Title: Efficacy and Tolerability Study of Device, RD047-26 for the Treatment of Mild to Moderate Atopic Dermatitis in Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oculus Innovative Sciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MIC-AD-001
Record Dates: First submitted 2010-10-26; First posted 2010-11-02 (Estimated); Last update posted 2012-05-30 (Estimated); Status verified 2012-05

CONDITIONS: Atopic Dermatitis; Pruritus
Keywords: Atopic Dermatitis; Pruritus
MeSH Terms: conditions — Dermatitis, Atopic; Pruritus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- RD047-26 (Experimental): Study Device
  Interventions: Device: RD047-26

INTERVENTIONS:
Device: RD047-26 — RD047-26 emollient gel

SUMMARY:
The purpose of this study is to find out if investigational device, RD047-26, is safe and useful for the treatment of mild to moderate atopic dermatitis.

DETAILED DESCRIPTION:
RD047-26, a device, may be tolerable and effective for the treatment of mild to moderate atopic dermatitis with associated pruritus in adults. The treatment effect will be evaluated by the subject and investigator.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Female or male, 18 to 65 years of age and in good general health
* Clinical diagnosis of stable mild to moderate atopic dermatitis
* Willing and able to follow study instructions and likely to complete all study requirements

Exclusion Criteria:

* Severe or uncontrolled asthma
* Pregnant, nursing, or planning a pregnancy during the study; or is a WOCBP but is not willing to use an effective method of birth control
* Current enrollment in an investigational drug or device study or participation in such a study within the last 30 days prior to Baseline (Day 0)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2010-10; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Investigator Global Assessment | 2 weeks
  Investigator Global Assessment of Atopic Dermatitis Severity

SECONDARY OUTCOMES:
Investigator Pruritus Assessment | 2 weeks
  Investigator Pruritus Severity Assessment
Subject Itch Assessment | 2 weeks
  Subject assessment of itch severity
Adverse Events | 2 weeks
  Number of subjects with related adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Zoe Draelos, M.D., Principal Investigator — Dermatology Consulting Services, High Point NC
Locations (1):
- Dermatology Consulting Services, High Point, North Carolina, United States